CLINICAL TRIAL: NCT01758185
Title: Phase 4 Safety and Immunogenicity Study of Aleph Inactivated Split Influenza Vaccine
Brief Title: Safety and Immunogenicity Study of Aleph Inactivated Split Influenza Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BJCDPC-3
Record Dates: First submitted 2012-12-20; First posted 2013-01-01 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2013-03

CONDITIONS: Healthy
Keywords: Inactivated split influenza vaccine; Immunogenicity; Safety; Consistence
MeSH Terms: interventions — Hepatitis B Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- recombinant hepatitis b vaccine (Placebo Comparator): 0.5ml intramuscular
  Interventions: Biological: recombinant hepatitis b vaccine; Biological: Aleph influenza vaccine
- Aleph influenza vaccine (Experimental): 0.5ml intramuscular
  Interventions: Biological: recombinant hepatitis b vaccine; Biological: Aleph influenza vaccine

INTERVENTIONS:
Biological: recombinant hepatitis b vaccine — 0.5ml intramuscular
Biological: Aleph influenza vaccine — 0.5ml intramuscular

SUMMARY:
The objective of this study was to evaluate the safety and immunogenicity of one inactivated split influenza vaccine, a primarily Chinese-marketed trivalent vaccine.

DETAILED DESCRIPTION:
A total of 3308 subjects were stratified equally into four age groups and receive either influenza vaccine or recombinant hepatitis b vaccine (seen as placebo). Systematic and local adverse reactions were reported for 28 d after the vaccination. Antibody levels were detected through hemagglutination inhibition assay before vaccination (Baseline) and 28d after the vaccination.

ELIGIBILITY:
Inclusion Criteria:

* more than three years in good healthy

Exclusion Criteria:

* current infectious fever or acute disease
* upper respiratory infectious symptom within 6m
* a history of allergy
* laboratory confirmed influenza
* autoimmune disease
* have get influenza vaccine since 2008

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3308 (Actual)
Dates: Start 2011-08; Primary Completion 2011-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Incidence rate of adverse events of the inactivated split influenza vaccine | two years

SECONDARY OUTCOMES:
Antibody titre of the inactivated split influenza vaccine | two years

CONTACTS AND LOCATIONS:
Overall Officials: Nianmin Shi, Master, Principal Investigator — Beijing Chaoyang District Center for Disease Control and Prevention
Locations (2):
- China (2):
  - Xinglong County Center for Disease Control and Prevention, Zhangjiakou, Hebei
  - Zhuolu County Center for Disease Control and Prevention, Zhangjiakou, Hebei

REFERENCES:
- [Derived] Bai Y, Shi N, Lu Q, Yang L, Wang Z, Li L, Han H, Zheng D, Luo F, Zhang Z, Ai X. Immunological persistence of a seasonal influenza vaccine in people more than 3 years old. Hum Vaccin Immunother. 2015;11(7):1648-53. doi: 10.1080/21645515.2015.1037998. PMID 26083828
- [Derived] Li S, Li L, Ai X, Yang L, Bai Y, Wang Z, Han H, Lu Q, Luo F, Zhang Z, Liu C, Xiao J, Shi N. A randomized, controlled, blinded study of the safety, immunogenicity and batch consistency of Aleph inactivated split influenza vaccine made in China in Chinese people. Hum Vaccin Immunother. 2014;10(3):557-65. doi: 10.4161/hv.27329. Epub 2013 Dec 3. PMID 24301228